CLINICAL TRIAL: NCT01335815
Title: High Sensitive Troponin T (hsTnT) and Copeptin as Prognostic Parameters in Patients With Elective Knee and Hip Endoprosthesis
Brief Title: High Sensitive Troponin T (hsTnT) and Copeptin as Prognostic Parameters in Patients With Elective Total Endoprosthesis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Prof. Dr. Evangelos Giannitsis, Department of Cardiology, University of Heidelberg
Other Study IDs: TnT hs 3
Record Dates: First submitted 2011-04-13; First posted 2011-04-14 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: Perioperative Myocardial Infarctions; Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — normal lab parameters
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- elective knee and limb endoprothesis

SUMMARY:
Summary: The purpose of the study is to prove if the biomarker high sensitive troponin T (hsTnT) and the biomarker of endogenous stress copeptin can serve as surrogate parameter of prognosis in patients with elective knee and hip total endoprosthesis.

DETAILED DESCRIPTION:
Consecutively, high sensitive troponin T and copeptin will be measured in all patients with elective knee and hip endoprosthesis in the orthopedic department of the University of Heidelberg. The blood is taken during the routine blood testes if possible, on admission and the days 1-4 following the operation. Usual baseline characteristics are taken as well as usual blood results (hb, cholesterol and so on). Primary endpoint is the detection of perioperative myocardial infarction and pulmonary embolism.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with elective knee and hip endoprosthesis

Exclusion Criteria:

* Not willing or not able to take part in the observational trial
* No written inform consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all patients with elective knee and hip endoprothesis
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Prevalence of perioperative myocardial infarction and pulmonary embolism | Until 96h after operation

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Giannitsis, Prof. Dr., Principal Investigator — Heidelberg University
Locations (1):
- University of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany